CLINICAL TRIAL: NCT04954950
Title: An Epidemiological Study on Winter Sports Injury in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019456
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Sports Injury
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sports injuries: Patients were classified according to self-reported years of participation in skiing and snowboarding: beginner (first season), medium (1-5 years), advanced (5-10 years) and expert (≥10 years). Date of injury was divided into weekdays and weekends/ holidays according to the Chinese government holiday arrangement.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aims of the study are to describe the injury patterns among recreational skiers and snowboarders in China and to provide primary data to guide the reconstruction of regional healthcare facilities to deal with the increasing number of participants in snow sports.

DETAILED DESCRIPTION:
A retrospective study was performed in Ski Resorts in Chongli, China. 5000-10000 injured skiers and snowboarders will be recruited. Data of all injury patients in the resort clinic will be collected. Patients' information, including sex, age, equipment, skill level and injured body part, will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Skiing and snowboarding injuries

Exclusion Criteria:

* Skiing and snowboarding visitors without injuries

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Data for this retrospective study were collected from the resort clinic in Chongli during ski season. Chongli is a destination ski resort in Northern China which has various terrains and has the largest number of annual visits.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
sex | 1 week after injury
  male/female
age | 1 week after injury
  15-60/>60
Equipment | 1 week after injury
  Equipment was classified into skis and snow-boards. Special equipment such as cross-country skis and skiboards is rare in China and has not been recorded in the present study.
Skill level | 1 week after injury
  Patients were classified according to self-reported years of participation in skiing and snowboarding: beginner (first season), medium (1-5 years), advanced (5-10 years) and expert (≥10 years).
Date of injury | 1 week after injury
  Date of injury was divided into weekdays and weekends/holidays according to the Chinese government holiday arrangement.
Causes of injury | 1 week after injury
  We summarised causes of injury into two types according to the subjective description of the scene of injury: not involving others, defined as falling or crashing without any body contact with others; and involving others, defined as crashing that involves two or more people.
Slope difficulty | 1 week after injury
  Slope difficulty was categorised into beginner trail, medium trail and advanced trail according to the official data of slope inclination angle.
Injured body parts | 1 week after injury
  Injured body parts were categorised into the following four anatomical body regions: (1) head/cervical, (2) torso, (3) upper extremity and (4) lower extremity.

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided